CLINICAL TRIAL: NCT03920228
Title: A Multicenter, Four-Part, Phase 2/3 Study Evaluating the Safety and Efficacy of PTX-022 in the Treatment of Adults With Moderate to Severe Pachyonychia Congenita
Brief Title: Phase 2/3 Study Evaluating the Safety and Efficacy of PTX-022 in Treatment of Adults With Pachyonychia Congenita
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PALV-02
Record Dates: First submitted 2019-04-02; First posted 2019-04-18 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Pachyonychia Congenita
Keywords: PC
MeSH Terms: conditions — Pachyonychia Congenita

STUDY DESIGN:
Intervention Model Description: This study consists of 2 treatment periods:
  * Open-Label
  * Randomized, Double-Blind, Placebo controlled
Who Masked: Participant, Investigator
Masking Description: During the open-label period, there is no masking. During the randomized, double-blind, placebo-controlled period the participant and Investigator are masked.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Open label period (Experimental)
  Interventions: Drug: PTX-022
- Randomized period - Dosing A (Placebo Comparator)
  Interventions: Drug: Placebo
- Randomized period - Dosing B (Experimental)
  Interventions: Drug: PTX-022; Drug: Placebo
- Randomized period - Dosing C (Experimental)
  Interventions: Drug: PTX-022

INTERVENTIONS:
Drug: PTX-022 — PTX-022 QTORIN
  Arms: Open label period; Randomized period - Dosing B; Randomized period - Dosing C
Drug: Placebo — Placebo topical
  Arms: Randomized period - Dosing A; Randomized period - Dosing B

SUMMARY:
This study evaluates the safety and efficacy of PTX-022, topical rapamycin, in the treatment of adults with moderate to severe Pachyonychia Congenita.

This study includes four-parts, and if a participant completes all parts, the participant will have received at least 3-months of PTX-022 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years or older
* Diagnosed Pachyonychia Congenita (PC), genetically confirmed
* Moderate to Severe PC
* Able and willing to comply with all protocol-required activities
* Willing and able to provide written informed consent

Exclusion Criteria:

* Any significant concurrent condition (including involving the inferior to the ankle) that could adversely affect participation.
* Any intentional changes in the patient's daily activities (associated with standing, walking and keeping balance), not resulting from an improvement in the patient's condition due to treatment.
* Patient's deemed by the investigator as unwilling or unable to remain compliant with all tests and procedures, including adherence to study drug administration and other protocol-required activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Patient Global Assessment of Activities Scale | 6 months

SECONDARY OUTCOMES:
Clinician Global Impression of Change Scale | 6 months
Pain at its worst as assessed by numerical rating scale | 6 months
Number of steps taken as assessed by activity monitor | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Hansen, MD, Principal Investigator — University of Utah; Joyce Teng, MD, Principal Investigator — Stanford University
Locations (9):
- United States (9):
  - Arizona Research Center, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - International Dermatology Research, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - Paddington Testing Co., Philadelphia, Pennsylvania
  - University of Utah, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PC Project — https://www.pachyonychia.org/
- See also: Palvella Therapeutics, Inc. — http://www.palvellatx.com